CLINICAL TRIAL: NCT03753126
Title: Leaflet Thickening and Stent Geometry in Sutureless Bioprosthetic Aortic Valves
Brief Title: Stent Geometry in Sutureless Bioprosthetic Valves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Magnus Dalén, MD PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: Perceval Geometry
Record Dates: First submitted 2018-11-22; First posted 2018-11-26 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Aortic Valve Stenosis; Heart Valve Diseases
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

ARMS (1):
- Cardiac CT imaging (Other)
  Interventions: Radiation: 4-dimensional volume-rendered computed tomography

INTERVENTIONS:
Radiation: 4-dimensional volume-rendered computed tomography

SUMMARY:
A single-center prospective interventional trial. Patients implanted with a sutureless bioprosthetic aortic valve at Karolinska University Hospital in Stockholm, Sweden from 2012 will be eligible. 4-dimensional volume-rendered computed tomography (CT) of the heart will be performed. The aim of the CT is to assess valve geometry and hypo-atrenuated leaflet thickening. Results of the CT examination, preoperative clinical characteristics, and postoperative clinical data will be registered. Data will be collected prospectively and retrospectively. Informed consent will be obtained from patients meeting the inclusion criteria before the initiation of any study-specific procedures.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a sutureless Perceval (LivaNova) sutureless bioprosthetic aortic valve at Karolinska University Hospital in Stockholm, Sweden between 2012 and 2016
* Provide written informed consent

Exclusion Criteria:

•Contraindication for CT with intravenous contrast injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Regional expansion of valve prosthesis | At CT performed once no less than 30 days and up to 10 years after aortic valve replacement
  Regional expansion measured using the angle formed by the border of each prosthetic leaflet and the centre point of the valve
Overall expansion of valve prosthesis | At CT performed once no less than 30 days and up to 10 years after aortic valve replacement
  Overall expansion of the implanted prosthesis calculated as the ratio between the ex vivo cross-sectional area and the in vitro cross-sectional area of the implanted valve

SECONDARY OUTCOMES:
Eccentricity of valve prosthesis | At CT performed once no less than 30 days and up to 10 years after aortic valve replacement
  Eccentricity of the implanted prosthesis calculated as ([max diameter-min diameter]/max diameter)×100

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Dalén, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Themudo R, Kastengren M, Bacsovics Brolin E, Cederlund K, Svensson A, Dalen M. Leaflet thickening and stent geometry in sutureless bioprosthetic aortic valves. Heart Vessels. 2020 Jun;35(6):868-875. doi: 10.1007/s00380-020-01553-9. Epub 2020 Jan 16. PMID 31950251